CLINICAL TRIAL: NCT04232605
Title: Investigation of Vasodilation and Intensity of Headache Triggered by Glucagon-like Peptide-1 in Healthy Volunteers and Migraine Patients
Brief Title: Investigation of Vasodilation and Intensity of Headache Triggered by Glucagon Like Peptide-1 in Humans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Hashmat Ghanizada, Principal investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: H-19037051
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — glucagon-like peptide 1 (7-37)-proline, glycyl(2)-

STUDY DESIGN:
Intervention Model Description: Phase one: In a randomized, single-blind, multiple-ascending-dose finding pilot study we investigate the safety and tolerability of GLP-1 on three healthy volunteers. The following GLP-1 doses will be given intravenously ( 1.5, 2.0 and 2.5 picomol/kg/min) over 20 min. The dose with considerable dilatory effect will be chosen for main study.
  Phase 2 and 3:The study is a double-blinded, placebo-controlled, randomized crossover study. It involves two arms, GLP-1 and placebo. Each participant will in a randomized order receive placebo or GLP-1 intravenous infusion over 20 min on the two experiment days.
  The study consists of two separate substudies, one for healthy volunteers and one for migraine patients. The substudies are otherwise identical.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GLP-1 (Active Comparator): Receive intravenous infusion of GLP-1.
  Interventions: Other: GLP-1 peptide
- Placebo (Placebo Comparator): Receive intravenous infusion of saline.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: GLP-1 peptide — Receive intravenous infusion of GLP-1. The dosage will be determined after a dose finding pilot study.
  Arms: GLP-1
Other: Placebo — Receive intravenous infusion saline
  Arms: Placebo

SUMMARY:
Studying glucagon-like peptide-1 (GLP-1) induced vasodilatory effects on extra - and intracerebral arteries and headache in healthy volunteers and migraine patients without aura.

DETAILED DESCRIPTION:
The purpose of this study is to examine the association between vasodilation and intensity of headache triggered by glucagon-like peptide 1 (GLP-1) in healthy volunteers and migraine patients without aura.

ELIGIBILITY:
Criteria for the healthy volunteers group

Inclusion Criteria:

* Healthy men/women.
* Age 18 to 60 years old.
* Weight 50 to 100 kg.

Exclusion Criteria:

* Tension headache more than 5 days a month in the preceding year.
* All other primary headache types.
* Headache on the examination day or within 48 hours before infusion of the study drug.
* Smoking.
* Daily intake of medicine of any kind except for peroral contraceptives.
* Women, who on the day of examination is 2 days before or 3 days from the first day of bleeding.
* Hypertension or hypotension.
* Coronary heart disease of any kind, as well as cerebrovascular disease.
* Pulmonary disease.
* Allergy to contents in the study drug.
* Psychiatric disease or substance abuse.
* Disease of any kind which the examining doctor deems relevant for participation in the study.
* Renouncing the right to information concerning own health.

Criteria for the migraine patients group

Inclusion Criteria:

* Migraine patients, who fulfill the ICHD-3 criteria for migraine without aura.
* Age 18 to 60 years old.
* Weight 50 to 100 kg.

Exclusion Criteria:

* Tension headache more than 5 days a month in the preceding year.
* All other primary headache types.
* Headache on the examination day or within 48 hours before infusion of the study drug.
* Smoking.
* Daily intake of medicine of any kind except for peroral contraceptives.
* Women, who on the day of examination is 2 days before or 3 days from the first day of bleeding.
* Hypertension or hypotension.
* Coronary heart disease of any kind, as well as cerebrovascular disease.
* Pulmonary disease.
* Allergy to contents in the study drug.
* Psychiatric disease or substance abuse.
* Disease of any kind which the examining doctor deems relevant for participation in the study.
* Renouncing the right to information concerning own health.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Vasodilation | 120 minutes
  Difference in circumference (in millimeter) of intra - and extracranial blood vessels before and after GLP-1 or placebo infusion, measured by transcranial doppler and ultrasound (Derma scan) at 10 specific time points (-10, 10, 20, 30, 40, 50, 60, 80, 100, and 120 minutes)
Headache intensity | 12 hours
  Headache intensity will be measured using Numerical rating scale (NRS) from ( 0 to 10 )

SECONDARY OUTCOMES:
blood pressure | 120 minutes
  Blood pressure (systolic and diastolic) in mmhg will be measured every 10 minutes
Facial skin perfusion | 120 minutes
  Non-invasive measuring of facial skin perfusion by laser speckle contrast imager.
Heart rate | 120 minutes
  heart rate will be measured every 10 minutes
Plasma glucose | 120 minutes
  Plasma glucose will be measured using (mmol/L) a ABL Radiometer, Denmark Blood-gas analyser

CONTACTS AND LOCATIONS:
Locations (1):
- Dansk Hovedpinecenter, Glostrup Municipality, Denmark